CLINICAL TRIAL: NCT07190950
Title: Effects of Low-level Laser Therapy on Soft and Hard Tissue Healing After Impacted Mandibular Third Molar Extraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Hoang Ngoc Hiep, DDS. Nguyen Hoang Ngoc Hiep, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24368-ĐHYD
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Third Molars Extraction; Low Level Laser Therapy; Bone Healing
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): After had third molar extraction at one side, patients do not receive low level laser therapy at this site (by not activating the tip)
- Experiment arm (Experimental): After had third molar extraction at the other side, patients receive 7 sessions of low level laser therapy at this side (the day of surgery, then first day, third day, seventh day, fourteenth day, twenty first day, twenty eighth day after surgery)
  Interventions: Procedure: Low Level Laser Therapy

INTERVENTIONS:
Procedure: Low Level Laser Therapy — Patients will receive LLLT at one side after third molar extraction surgery. There will be 7 sessions at the day of surgery, then first, third, seventh, fourteenth, twenty first, twenty eighth day after surgery.
  Other Names: LLLT
  Arms: Experiment arm

SUMMARY:
Impacted lower third molar extraction is one of the most commonly performed dental procedures in daily practice. However, this is considered a relatively invasive procedure. During the surgery, dental surgeon must reflect a full-thickness flap, remove bone to expose the tooth, section and deliver the tooth. As a result, after surgery, patients often experience many complications, from swelling, pain, jaw tightness, etc. to alveolar bone loss, periodontal problems distal to the second molar, etc.

Therefore, clinicians are always looking for additional therapies to minimize complications, helping patients have a more comfortable experience after wisdom tooth surgery.

To date, placing grafting materials such as bone or other biological materials (growth factors, platelet-rich plasma, platelet-rich fibrin) into the tooth socket has been shown to be able to preserve the alveolar crest after extraction. However, these materials require preparation time, are costly, and have the risk of infection related to bone grafts.

Meanwhile, low-level laser therapy (LLLT) is known as a safe, non-invasive therapy that can affect cell metabolism without causing tissue damage. This therapy has been widely applied in many fields of medicine in general and in dentistry in particular. Low-level lasers have been studied to help reduce swelling, pain, and jaw tightness after impacted lower wisdom teeth surgery. In vitro or in vivo studies evaluating the healing effect of low-level lasers have given very positive results. However, there is still a lack of scientific evidence to prove the healing effect of low-level lasers on human tooth extraction sockets.

The study we conducted is a scientific study, in the field of Dentistry. This study aimed to evaluate the effectiveness of low-level laser on soft tissue and bone healing after surgical extraction of impacted lower third molars in a group of Vietnamese population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (at least 18 years of age) have both jaws lower impacted third molars indicated to be extracted. Both teeth are the same of

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
wound healing score | at third, seventh and thirtieth day after third molar extraction surgery
  Base on IPR scale (Inflammatory Proliferative Remodeling Scale) by Hamzani et al. (2018)
New bone density | The day of surgery, first and third month after surgery
  Based on periapical X-rays taken on the day of surgery right after extraction, first and third month, we calculate new bone density by calculate the pixel density at extracted socket.
Changing of alveolar crest level distal to second lower molar | the day of surgery, first and third month after third molar extraction surgery
  After taking periapical X-rays on the day of surgery right after extraction, first and third month, we measure alveolar crest level distal to second lower molar from the base of extracted socket to cemento-enamel junction (CEJ) of second molar (the reference is a 5 mm stainless steel straight wire buried in rubber impression)

CONTACTS AND LOCATIONS:
Overall Officials: Ly Thi Bich Nguyen, Doctor of Philosophy, Study Director
Locations (1):
- University of medicine and pharmacy at Ho Chi Minh city, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided